CLINICAL TRIAL: NCT06986330
Title: Endovascular Treatment of Cerebrovascular Diseases Guided by Optical Coherence Tomography (OCT) Technology: a Prospective Observational Study （CVD-OCT） Subject Hosting Organization: The First Affiliated Hospital of Wannan Medical College (Yijishan Hospital) Principal Investigator: Xianjun Huang
Brief Title: Endovascular Treatment of Cerebrovascular Diseases Guided by Optical Coherence Tomography (OCT) Technology（CVD-OCT）
Acronym: （CVD-OCT)
Status: Active, not recruiting | Type: Observational
Sponsor: First Affiliated Hospital of Wannan Medical College (Other)
Responsible Party: Sponsor
Other Study IDs: 20231130
Record Dates: First submitted 2025-05-15; First posted 2025-05-23 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Carotid Stenosis; Optical Coherence Tomography (OCT); Endovascular Treatment
MeSH Terms: conditions — Carotid Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- oct: The diagnosis and treatment behavior of all subjects in this study followed the requirements of the current guidelines, and there were no additional interventions.

SUMMARY:
OCT techniques have been used in the assessment of both intracranial and extracranial lesions.(1) Preprocedural evaluation: The morphologic characteristics of carotid atherosclerotic plaques can be evaluated by OCT before surgery to identify vulnerable plaques and guide interventional therapy. It has been shown that plaque image features observed by OCT and based on the "thin fibrous cap" characteristics of plaques can predict rupture and thrombotic risk of atherosclerotic plaques. Similarly, the results of studies based on OCT plaque features suggest that OCT plaque features can be used for the identification of symptomatic carotid plaques.The results of studies based on OCT plaque characteristics suggest that OCT plaque characteristics correlate with the degree of carotid stenosis and ischemic symptoms. Therefore, it is important to use OCT to assess plaque characteristics prior to cerebrovascular interventions and to identify high-risk plaques that are prone to cause ischemic events, in order to guide carotid interventions, especially for patients whose stenosis has not reached the level of intervention, but who have not yet reached the level of ischemic events, or who are at risk of ischemic events.lesions with stenosis not reaching the level of intervention but with the presence of vulnerable plaques are of great significance.(2) Evaluation of immediate post-interventional outcomes: Currently, OCT has been used to evaluate the expansion rate of the relevant stent immediately after stenting, stent adherence, protrusion of diseased tissue into the lumen of the vessel, and in-stent thrombosis.In addition, in acute occlusion recanalization of intracranial vessels, the application of OCT can identify the nature of lesions during treatment, such as clips, atherosclerotic stenosis, and other lesions, and guide the development of surgical strategies. (3) Interventional follow-up: OCT can be used in post-interventional follow-up for post-stenting endothelial repair, in-stent restenosis, de novo atherosclerosis, and thrombus formation.

In summary, OCT can accurately assess the nature of cerebrovascular lesions and plaques and guide clinical interventions.For medical centers that have the conditions, it is recommended to standardize the application of OCT to guide the interventional precision treatment of ischemic cerebrovascular disease.In the future, a clinical study database of OCT in Chinese patients with ischemic cerebrovascular disease should be established to provide evidence-based medical evidence of OCT in the diagnosis and treatment

DETAILED DESCRIPTION:
Stroke is a kind of acute focal damage to the central nervous system caused by vascular lesions, resulting in neurological function defects. With the characteristics of high morbidity, high disability rate and high mortality rate in the world, it has become the second largest cause of death in the world and the first fatal and disable disease in China 1. A national epidemiological survey of stroke in China (NESS-China) shows that about 1,596 people per 100,000 people in China have been diagnosed For stroke, the age-standardized prevalence and incidence of stroke are 1,115/100,000 and 247/100,000 years 2. Stroke has brought a huge burden of disease to the residents of China. How to prevent and treat stroke is a major task in China's health industry.

1.1 Ischemic stroke and atherosclerosis

Stroke is divided into ischemic stroke and hemorrhagic stroke, of which ischemic stroke accounts for 80%. The etiology of ischemic stroke can be divided into aortic atherosclerosis type (Large-at) according to the trial of Org 10172 in Acute Stroke Treatment (TOAST) Ery atherosclerosis, LAA), cardiogenic embolism type, small arterial occlusion type, other causal type and unexplained type 5 types 3. LAA-type ischemic stroke refers to the stenosis or occlusion of more than 50% of the main trunk or cortical branches of the cerebrovascular caused by atherosclerosis, resulting in the symptoms of the corresponding blood supply area. A number of studies based on Chinese hospital data show that the proportion of LAA ischemic stroke varies from region to region, ranging from 11.4% to 67.6% 4. On the surface of the study, about 30%-50% of ischemic stroke can be attributed to intracranial atherosclerotic stenosis, and about 8%-10% of ischemic stroke can be attributed to carotid atherosclerosis.

The occurrence, development and complications of atherosclerosis is a slow process. It is a chronic inflammatory reaction of vascular endothelial cell dysfunction combined with macrophages, smooth muscle cells and low-density lipoprotein cholesterol, as well as a variety of inflammatory factors, which can lead to endovascular lipid deposition and fibrous proliferation. , calcium sedimentation, cholesterol crystallization, plaque erosion, plaque rupture, thrombosis; medium membrane thinning, fiber proliferation; a series of slow-progressing pathophysiological processes with narrowing and even occlusion of the lumen 6. As a common cause of ischemic stroke, the pathophysiological mechanism of ischemic stroke is divided into 2 categories: 1 The formation of atherosclerotic plaques of large blood vessels inside and outside the skull leads to severe narrowing or even occlusion of the lumen, resulting in reduced perfusion of brain tissue and ischemic infarction; 2 The thrombus on the surface of large vascular plaques can be shed with blood flow. It causes distal vascular embolism, causing ischemic infarction of brain tissue in the corresponding blood supply area.

1.2 Diagnosis and treatment strategies and dilemmas of cerebral vascular atherosclerotic stenosis

At present, the treatment of patients with cerebral vascular atherosclerotic stenosis mainly includes drug treatment and surgical treatment or intravascular intervention treatment. Drug treatment includes anti-platelet aggregation treatment and lipid regulation and plaque stabilization treatment. In addition, it also includes treatments such as risk factor control.

Surgical treatment or intravascular treatment: A number of randomized controlled studies have shown that symptomatic carotid artery patients with stenosis degree of ≥50% diagnosed by transcerebrovascular digital subtraction angiography (DSA) and patients with asymptomatic carotid stenosis with stenosis degree of ≥70%, carotid endatrial stripping or carotid branch can be adopted. Frame implantation is used to reduce the risk of stroke or recurrence. 9,10 For patients with unfavorable anatomical structure of the neck, stenosis after carotid inner membrane peeling, accompanied by perioperative risk, previous radiotherapy history or other patients who can increase the risk of endometrial stripping, less invasive carotid stent implantation can be used for treatment.

The evidence-based evidence is still insufficient for the superiority and inferiority of the efficacy of intravascular interventional treatment in patients with intracranial artery stenosis and the efficacy of the best drug treatment. Current studies show that intravascular interventional treatment has failed to reduce the risk of stroke recurrence in patients with symptomatic intracranial atherosclerotic stenosis compared with simple drug treatment, which may be related to the screening of patients. Previous randomized controlled trials screened patients only based on the degree of stenosis of the vascular lumen, ignoring the impact of plaque characteristics on the risk of stroke. More and more evidence shows that the risk of stroke is closely related to plaque vulnerability.

Although DSA is currently the gold standard for the diagnosis of cerebral vascular stenosis, DSA cannot recognize plaque characteristics. In recent years, with the development of vascular wall imaging technology, more and more research on plaque susceptibility and stroke risk have become more and more profound. These studies may change the treatment strategy of patients with cerebral atherosclerosis.

1.3 Application of optical coherence tomography (OCT) technology in cerebral vascular atherosclerotic stenosis

OCT technology is used in the evaluation of intracranial and extracranial lesions. ( 1) Preoperative evaluation: The morphological characteristics of carotid atherosclerotic plaques can be evaluated through OCT before operation, so as to identify vulnerable plaques and guide interventional treatment. Studies have shown that through the plaque image characteristics observed by OCT and based on the "thin fiber cap" characteristics of the plaque, the rupture of atherosclerotic plaque and the risk of thrombosis can be predicted, and symptomatic carotid plaques can be identified. Similarly, the research results based on the characteristics of OCT plaque show that there is a certain correlation between the characteristics of OCT plaque and the degree of carotid artery stenosis and ischemic symptoms. Therefore, it is important to use OCT to evaluate the characteristics of plaques before cerebrovascular interventional treatment, identify high-risk plaques that are prone to ischemia events, and guide carotid interventional treatment, especially for lesions where the degree of vascular stenosis does not reach the level of intervention, but there are susceptible plaques. ( 2) Evaluation of the immediate effect after interventional treatment: At present, OCT has been used to evaluate the immediate expansion rate of the relevant stent after stent placement, stent wall adhession, the protrusion of lesion tissue into the vascular cavity and thrombosis in the stent, etc. In addition, in intracranial vascular acute occlusion and re-permission surgery, the application of OCT can identify the nature of lesions in the treatment process, such as dissection, atherosclerotic stenosis and other lesions, and guide the formulation of surgical strategies. ( 3) Interventional treatment follow-up: OCT can be used for follow-up after interventional treatment to understand the repair of the inner membrane after stent, stent re-stenosis, neonatal atherosclerosis and thrombosis, etc.

In summary, OCT can accurately evaluate the nature of cerebrovascular lesions and plaques, and guide clinical interventional diagnosis and treatment. For qualified medical centers, it is recommended to apply OCT in a standardized way to guide the interventional and accurate treatment of ischemic cerebrovascular disease. In the future, an OCT clinical research database for patients with ischemic cerebrovascular disease in China should be established to provide evidence-based medical evidence of OCT in the diagnosis and treatment of cerebrovascular disease.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of cerebrovascular disease (including asymptomatic patients);
2. Cerebral angiography or intervention with OCT is required in the course of clinical diagnosis and treatment;
3. Informed consent signed by the patient or the patient's legally authorized representative.

Exclusion Criteria:

1. Patients with contrast allergy or intolerance to iodine contrast;
2. Patients with tortuous blood vessels who are unable to complete OCT.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Visiting Yijishan Hospital and needing endovascular treatment for carotid artery stenosis
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-11-30 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Main study outcomes | Before and 3 days after surgery
  Evaluation of the characteristics of lesions in various types of cerebrovascular diseases. Use of high-resolution magnetic resonance to compare changes in different sequences of patients preoperatively and postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Wannan Medical College, Wuhu, Anhui, China

IPD SHARING:
Plan to Share IPD: Yes